CLINICAL TRIAL: NCT06848842
Title: A Phase II Clinical Study of Ivonescimab Plus CAPOX Regimen in Patients With Initially Unresectable Colorectal Cancer Liver-only Metastases
Brief Title: Ivonescimab Plus Chemotherapy in Patients With Initially Unresectable Colorectal Cancer Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5043
Record Dates: First submitted 2025-02-06; First posted 2025-02-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal Liver Metastases; initially unresectable; ivonescimab; objective response rate
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Ivonescimab plus chemotherapy
  Interventions: Drug: Ivonescimab plus chemotherapy

INTERVENTIONS:
Drug: Ivonescimab plus chemotherapy — Ivonescimab, 20mg/kg, D1, Q3W; Oxaliplatin, 130mg/m2, D1, Q3W; Capecitabine, 1000mg/m2, BID, D1-D14, Q3W

SUMMARY:
The goal of this clinical trial is to learn if ivonescimab plus chemotherapy works to treat colorectal cancer liver metastases that cannot be completely removed. It will also learn about the safety of ivonescimab. The main questions it aims to answer are:

Does ivonescimab plus chemotherapy raise the objective response rate? What medical problems do participants have when receiving ivonescimab plus chemotherapy?

Participants will:

Receive ivonescimab and chemotherapy every 3 weeks, no more than 8 cycles. Visit the clinic once every 2 cycles (6 weeks) for checkups and tests. Receive curative surgery, maintenance therapy, or discontinue study treatment according to the expert team's evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically confirmed colorectal adenocarcinoma.
3. Radiologically confirmed liver-only metastases. Patients with ≤1 cm extrahepatic lesions not confirmed as metastatic are eligible.
4. No prior systemic therapy or local therapy for metastatic lesions, or completion of neoadjuvant/adjuvant chemotherapy ≥6 months before diagnosed disease recurrence.
5. Liver metastases considered unresectable or borderline resectable by multidisciplinary evaluation.
6. Liver metastases were measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. Eastern Cooperative Oncology Group performance status 0-1
8. Life expectancy ≥12 weeks.
9. No contraindications to hepatic resection/ablation, and primary tumor resectable or previously resected.
10. Adequate organ function as determined by normal bone marrow function (hemoglobin ≥80 g/L, absolute neutrophil count ≥1.5×10⁹/L, and platelets ≥100×10⁹/L), renal function (serum creatinine ≤1.5×upper limit of normal [ULN] and creatinine clearance ≥30 mL/min), liver function (serum bilirubin ≤2×ULN and serum transaminases ≤5×ULN).

Exclusion Criteria:

1. Definite extrahepatic metastases.
2. dMMR or MSI-H colorectal cancer.
3. Intolerance to the study drug during prior neoadjuvant/adjuvant therapy.
4. Toxicities from prior therapy have not resolved to ≤ Grade 1 (according to NCI-CTCAE v5.0), except for alopecia (any grade) and peripheral neuropathy (≤ Grade 2).
5. History of or concurrent other malignancies within the past 5 years, except cured localized tumors.
6. Surgery performed within 28 days prior to enrollment.
7. Hypertension with systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg despite antihypertensive treatment.
8. Major cardiovascular events within 12 months prior to enrollment.
9. History of severe bleeding tendency or coagulation disorders; tumor encasement of major blood vessels or significant necrosis or cavitation, and the investigator deems participation in the study may pose a bleeding risk.
10. Active autoimmune disease requiring systemic treatment within the past 2 years.
11. History of immunodeficiency, positive HIV antibody test, or long-term use of corticosteroids or other immunosuppressants.
12. Prior history of allogeneic bone marrow or organ transplantation.
13. Received live vaccines within 30 days prior to the first dose or plans to receive live vaccines during the study period.
14. Allergy to any component of the study drugs; history of severe hypersensitivity reactions to other monoclonal antibodies.
15. Women who are pregnant or breastfeeding.
16. Severe comorbidities or any other condition that precludes safe administration of the study treatment, including but not limited to symptomatic congestive heart failure (Class II or higher per NYHA classification), unstable angina, acute myocardial ischemia, poorly controlled arrhythmias, decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric/social conditions that may limit compliance with study requirements or impair the subject's ability to provide written informed consent.
17. Any other condition deemed by the investigator as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | At the end of Cycle 8 (each cycle is 21 days)
Treatment-Emergent Adverse Events | From the date of enrollment until 90 days after the Cycle 8 (each cycle is 21 days)

SECONDARY OUTCOMES:
No evidence of disease rate | 6 months
Progression-free survival | From date of enrollment until the date of first documented progression, assessed up to 2 years
Overall Survival | From date of enrollment until the date of death, assessed up to 2 years
Recurrence-free survival | From the date of curative resection until the date of first documented progression, assessed up to 2 years
Disease control rate | At the end of Cycle 8 (each cycle is 21 days)
Treatment-related adverse events | From the date of enrollment until 90 days after the Cycle 8 (each cycle is 21 days)
Immunotherapy-related adverse events | From the date of enrollment until 180 days after the Cycle 8 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No